CLINICAL TRIAL: NCT06176807
Title: Prediction of Acute Kidney Injury in Patients With Sepsis Using Venous Excess Ultrasound Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assistant professor, Mansoura University
Other Study IDs: MS.22.10.2155
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Intensive Care Unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Venous Excess Ultrasound Score — -- The IVC diameter : Grade 0: <5 mm with respiratory variation Grade I: 5-9 mm with respiratory variation Grade II: 10-19 mm with respiratory variation Grade III: >20 mm with respiratory variation Grade IV: >20 mm with minimal or no respiratory variation
  - Hepatic vein (HV) interrogation by pulsed wave Doppler identification and analysis of A, S, and D waves.
  Grade 0: normal S > D Grade I: S < D with antegrade S Grade III: S flat or inverted or biphasic trace - Portal vein Doppler (PD)as follow: Grade 0: <0.3 pulsatility index Grade I: 0.3-0.49 pulsatility index Grade III: 0.5-1.0 pulsatility index Pulsatility index is calculated as (Vmax - Vmin)/Vmax
  - VEXUS staging of venous congestion. (VEXUS ) Grade 0: IVC grade <III, HD grade 0, PV grade 0 Grade I: IVC grade IV, but normal HV/PV pattern Grade II: IVC grade IV with mild flow pattern abnormalities in HV/PV Grade III: IVC grade IV with severe flow pattern abnormalities in HV/PV

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. Sepsis and septic shock are major healthcare problems, killing between one in three and one in six of those they affect. organ dysfunction can be represented by the Sequential Organ Failure Assessment (SOFA) score of 2 points or more (respiratory rate of 22/min or greater, altered mentation, or systolic blood pressure of 100 mm Hg or less), which is associated with an in- hospital mortality greater than 10%.

Septic shock is defined as a subset of sepsis in which profound circulatory, cellular, and metabolic abnormalities are associated with a greater risk of mortality than with sepsis alone. Patients with septic shock can be clinically identified by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia. This combination is associated with hospital mortality rates greater than 40%.

DETAILED DESCRIPTION:
All patients with two out of four of Systemic Inflammatory Response Syndrome (SIRS) criteria (heart rate greater than 90, respiratory rate greater than 20, temperature greater or equal to 38 ⁰ C or less than 36⁰ C, altered mental state) and suspected infection and one of the following risk factors ( Age greater than 65 years, Recent surgery Immunocompromised AIDS, chemotherapy, neutropenia, diabetes, renal failure, hepatic failure, cancer, alcoholism)should be considered at risk of sepsis according to emergency department sepsis guidelines 2022.

The VExUS score ranges from Grades 0-3. In Grade 0, a non- dilated IVC (< 2 cm) indicates that no congestion is present. In Grades 1- 3, the IVC diameter is > 2 cm. In Grade 1, a dilated IVC and any combination of mildly abnormal flow patterns (but no severe features) indicates mild congestion. In Grade 2, a dilated IVC and one severely abnormal flow pattern indicates moderate congestion. In Grade 3, a dilated IVC and two or more severely abnormal flow patterns indicates severe congestion.

ELIGIBILITY:
Inclusion Criteria:

* All patients with sepsis.
* Patients aged between 21 and 65.
* Both sexes

Exclusion Criteria:

* Patients refused to participate in the study.
* Renal failure.
* Right ventricular dysfunction and dilatation.
* Moderate to severe tricuspid regurge.
* Cases of cirrhosis with liver cell failure.
* Inadequate window.
* IVC thrombus

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to evaluate combination of inferior vena cava diameter, hepatic venous flow, and portal vein pulsatility index: venous excess ultrasound score (VEXUS Score) in predicting acute kidney injury in patients with sepsis.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between serial VEXUS score and AKI in patients with sepsis. | 4 months
  Correlation between serial VEXUS score and AKI in patients with sepsis.

SECONDARY OUTCOMES:
Assess correlation between VEXUS score and hemodynamics: mean arterial pressure, central venous pressure, vasopressor use, urine output and daily fluid balance and serum lactate. | 4 months
  Assess correlation between VEXUS score and hemodynamics: mean arterial pressure, central venous pressure, vasopressor use, urine output and daily fluid balance and serum lactate.

CONTACTS AND LOCATIONS:
Locations (1):
- Nevert adel, Al Mansurah, Egypt